CLINICAL TRIAL: NCT00231920
Title: Prospective Pilot Safety Study Administering Two Doses of Inactivated Influenza Vaccine to Infants 10-22 Weeks of Age
Brief Title: Inactivated Influenza Vaccine in Infants 10-22 Weeks of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 04-057
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2006-11

CONDITIONS: Influenza
Keywords: Influenza, Vaccine, Infants
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

INTERVENTIONS:
Biological: Fluzone

SUMMARY:
This study proposes to enroll 50 young infants, ages 10 to 22 weeks. Each of the fifty infants will receive two 0.25mL doses of preservative-free Fluzone®, given a minimum of 28 days apart but no more than 42 days apart. Preservative-free Fluzone® will not be administered at the same time as other routine vaccines. Approximately 2-3mLs of blood sample will be obtained prior to the first vaccination, approximately 4 weeks after the second vaccination and 6 months after the second vaccination for the measurement of immune response. The primary purpose of this study is twofold: 1.) To determine the safety of administering two doses of preservative-free Fluzone® to young infants and 2.) To determine the capability of inducing an immune response of administering two doses of preservative-free Fluzone® to young infants.

DETAILED DESCRIPTION:
Influenza virus is an important global cause of morbidity and mortality. Influenza A or B viruses cause epidemics of disease almost every winter in the United States with an average of 36,000 deaths and 114,000 hospitalizations each year during 1990s (superscript 1). Children have the highest rates of infection while adults greater than 50 years of age have the highest mortality rates (superscript 2). Influenza, however, is associated with hospitalizations in young infants. In a survey of the Tennessee Medicaid database over many years, Neuzil et. al reported hospitalization rates in children less than 6 months of age that were much higher than in older children, and the rates approached those over 65 years of age (superscript 3). This is a prospective, phase l, open-label, self-contained, four visits over a period of 7 months, pilot study of 50 healthy infants, aged 10-22 weeks, with history of up-to-date routine immunizations, to assess safety and immunogenicity of administering 2 pediatric doses (with a minimum 4 weeks apart) of 0.25 ml of trivalent Influenza vaccine (Fluzone®). Each of the 50 infants will receive two 0.25mL doses of preservative free Fluzone®, given a minimum of 28 days apart but no more than 42 days apart. Preservative-free Fluzone® will not be administered at the same time as other routine vaccines. Approximately 2-3 mLs of venous blood will be obtained prior to the first vaccination, approximately 4 weeks after the second vaccination and 6 months after the second vaccination for the measurement of neutralization and HAI titers. Infants will be closely monitored during the influenza season for respiratory symptoms, fever, or other influenza-like illnesses. They will be seen during these episodes and nasal washes will be collected for a viral screen that will include culture for influenza virus, respiratory syncytial virus (RSV), adenovirus and parainfluenza virus and rapid test for influenza and RSV. Blood collected at the follow up visit, 6 months after the second dose of Fluzone®, will be used to measure post season antibody titers to strains of influenza A and B.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants, 10-22 weeks of age
2. Up to date with routine immunizations (Hepatitis B [Hep B]; diphtheria, tetanus and pertussis [DTaP]; pneumococci [Prevnar]; polio [IPV]; Haemophilus influenzae type B [Hib])
3. Free of obvious health problems as established by medical history and clinical examination before entering into the study
4. Parent/legal guardian willing and capable of signing written informed consent
5. Parent/legal guardian expected to be available for entire study
6. Parent/legal guardian can be reached by telephone.

Exclusion Criteria:

1. History of hypersensitivity to eggs or egg proteins
2. Former premature infants (<37 weeks)
3. History of wheezing or use of bronchodilator medication
4. History of hospitalization (excluding birth)
5. Significant underlying chronic illness (i.e. congenital heart defect, bronchopulmonary dysplasia, HIV)
6. Immunodeficiency disease or use of immunosuppressive therapy by the participant
7. Any other condition which in the clinical judgment of the investigator might interfere with vaccine evaluation
8. Current enrollment and participation in a clinical trial for an investigational drug or vaccine
9. Plans for participation in another clinical trial with an investigational drug or vaccine for the duration of this flu study.

Ages: 10 Weeks to 22 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2004-10; Primary Completion 2006-08 (Actual); Study Completion 2006-10

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee